CLINICAL TRIAL: NCT05237245
Title: Caractérisation Clinico- Biologique et Survie Des Patients Porteurs d'Une lymphoprolifération HTLV-1 Induite (ou Lymphome/leucémie lié au Virus HTLV-1) et Des Patients infectés Par le Virus HTLV-1
Brief Title: Clinico-biological Characterization and Survival of Patients With Adult T-cell Leukemia / Lymphoma (ATL) and Patients Chronically Infected With the HTLV-1 Virus (HTLV-OBS)
Acronym: HTLV-OBS
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP180684; 2020-A02320-39 (Other: ID-RCB Number)
Record Dates: First submitted 2021-12-20; First posted 2022-02-14 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Lymphoproliferation Induced by HTLV-1; HTLV-1 Adult T-cell Lymphoma / Leukemia; HTLV-1 Infection
Keywords: Human T-lymphotropic Virus 1; lymphoma; leukemia
MeSH Terms: conditions — Leukemia; HTLV-I Infections; Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, affected organ biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: Adult T-cell leukemia / lymphoma (ATL) patients
- 2: HTLV-1 chronically infected patients without ATL

SUMMARY:
The purpose of this study is to evaluate the outcome (survival) of Adult T-cell leukemia / lymphoma (ATL) patients who receive or not specific treatment for their hemopathy (cohort 1) and the outcome (survival) of HTLV-1 chronically infected patients with / without extra-haematological disorders (cohort 2).

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* HTLV-1 infected
* T lymphoproliferation induced by HTLV-1 (cohort 1)
* without T lymphoproliferation induced by HTLV-1 (cohort 2)
* informed and accepted the collection of data

Exclusion Criteria

- Patients refusal of participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with lymphoproliferation induced by HTLV-1 (or HTLV-1 adult T-cell lymphoma / leukemia) and HTLV-1 infected patients
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-03-23 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Number of survivors | Up to 1 year
  for cohorts 1 and 2

SECONDARY OUTCOMES:
Number of survivors at 2 years | At 2 years
  for cohorts 1 and 2
Number of survivors at 5 years | 5 years
  for cohorts 1 and 2
HTLV-1 proviral load | day 1
  for cohorts 1 and 2
viral integration profile | day 1
  for cohorts 1 and 2
lymphocyte phenotyping of tumor cells | day 1
  for cohorts 1 and 2
genetic analysis of tumor cells by Next-generation sequencing (NGS) | day 1
  for cohorts 1 and 2
number of patients with HTLV-1-related hematological disorders | day 1
  for cohort 1
number of patients with HTLV-1-related extra-hematological disorders | day 1
  for cohort 1
types of ATL | day 1
  According the Shimoyama classification (smoldering, chronic, Acute and Lymphoma) for cohort 1
Treatment lines | during 5 years
  Chemotherapy type, number of Chemotherapy cycles, efficacity of Chemotherapy : Number of complete remissions following treatment : for cohort 1
Response to induction therapy | during 5 years
  according to established response criteria for ATL for cohort 1
Progression free survival (PFS) | during 5 years
  for cohort 1
relapse-related mortality | during 5 years
  for cohort 1
chemotherapy-related mortality | during 5 years
  for cohort 1
transplant-related mortality | during 5 years
  for cohort 1
Number of serious adverse events according to WHO classification related to treatment received | during 5 years
  for cohort 1
Allograft-specific characteristic | during 5 years
  (donor type, conditioning type, engraftment, graft-related mortality) for cohort 1
number of progression to ATL | at 2 years
Number of progression to ATL | At 5 years
number of patients with HTLV-1-related extrahematological disorders | during 5 years
Number of patients with corticotherapy for extrahematological complications | during 5 years
  Dose of corticotherapy for extrahematological complications, number of days with corticotherapy for extrahematological complications
Number of Serious adverse events according to WHO classification related to treatment received | during 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Ambroise MARCAIS, MD, Principal Investigator — Assistance Publique-Hôpitaux Paris
Locations (1):
- Hôpital Necker Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No